CLINICAL TRIAL: NCT06301074
Title: A Multicenter, Randomized, Placebo-Controlled, Double-Blinded Phase Ⅰ Study to Evaluate the Tolerability and Pharmacokinetics of HS-10509 in Chinese Adult Subjects
Brief Title: The Phase I Study of HS-10509 in Chinese Adult Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HS-10509-101
Record Dates: First submitted 2024-02-26; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-02

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Psychotropic drugs; Antipsychotic agents
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Intervention Model Description: For each cohort, participants will be assigned to receive HS-10509 or placebo in parallel
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HS-10509 in healthy adults (Experimental): In SAD, participants in each dose-escalation cohort will orally receive a single dose of HS-10509 or a matching placebo on Day 1
  Interventions: Drug: HS-10509
- Placebo in healthy adults (Placebo Comparator): In SAD, participants in each dose-escalation cohort will orally receive a single dose of HS-10509 or a matching placebo on Day 1
  Interventions: Drug: Placebo
- HS-10509 in patients (Experimental): In MAD, patient with schizophrenia in each dose-escalation cohort will orally receive HS-10509 or a matching placebo once daily for 28 days.
  Interventions: Drug: HS-10509
- Placebo in patients (Placebo Comparator): In MAD, patient with schizophrenia in each dose-escalation cohort will orally receive HS-10509 or a matching placebo once daily for 28 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HS-10509 — In SAD, participants will be assigned to receive either HS-10509 or a matching placebo for a single administration. There are 5 predefined dose cohorts (each cohort including 8 for HS-10509 and 2 for placebo), initially starting at 10 mg for cohort 1.
  In MAD, participants will assigned to receive HS-10509 or a matching placebo once daily for 28 days. There will be 3 dose cohorts (each cohort including 8 for HS-10509 and 2 for placebo), and the dose for each cohort is to be determined.
  Arms: HS-10509 in healthy adults; HS-10509 in patients
Drug: Placebo — In SAD, participants will be assigned to receive either HS-10509 or a matching placebo for a single administration. There are 5 predefined dose cohorts (each cohort including 8 for HS-10509 and 2 for placebo), initially starting at 10 mg for cohort 1.
  In MAD, participants will assigned to receive HS-10509 or a matching placebo once daily for 28 days. There will be 3 dose cohorts (each cohort including 8 for HS-10509 and 2 for placebo), and the dose for each cohort is to be determined.
  Arms: Placebo in healthy adults; Placebo in patients

SUMMARY:
The study is to evaluate the safety, tolerability, and PK characteristics following single administration of HS-10509 in healthy adults, and multiple administrations of HS-10509 in patients with schizophrenia.

Participants will have HS-10509 tablets or placebo once in the single ascending dose (SAD) part or once daily for 28 days in the multiple ascending dose (MAD) part.

DETAILED DESCRIPTION:
This is a first-in-human, randomized, double-blinded, and placebo-controlled study.

In the single-ascending dose (SAD) part, subjects will receive HS-10509 tablets or placebo once. There are 5 predefined dose cohorts of 10 subjects each (including 8 for HS-10509 and 2 for placebo). SAD part of the study will assess the safety, tolerability, and PK characteristics of single ascending doses of HS-10509 to determine the dose range that is safe and well tolerated in healthy subjects.

In the multiple ascending dose (MAD) part, patients with schizophrenia will receive HS-10509 or placebo once daily for continously 28 days. There are 3 predefined dose cohorts with 10 subjects each (including eight for HS-10509 and 2 for placebo). MAD of the study will assess the safety, tolerability, PK and primary efficacy of multiple ascending doses of HS-10509 in subjects with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Part 1(SAD) for healthy adults

  1. When signing the ICF, the subject should be between 18 and 45 years old (inclusive);
  2. Have a full understanding of the trial content, process and possible adverse reactions, be willing and able to abide by the contraindications or restrictions stipulated in this program, and voluntarily sign the ICF;
  3. Male weight ≥50kg, female weight ≥45kg, body mass index (BMI= weight/height 2[kg/m2]) in the range of 18-28 (inclusive);
  4. Agree to use (or have their partner use) an effective contraceptive method from the date of signing the ICF until 90 days after the last dose, and there are no plans to donate eggs/sperm.
* Part 2 (MAD) for Schizophrenia patients

  1. When signing the ICF, the subject is between 18 and 65 years old (inclusive);
  2. BMI at screening and baseline was between 18.5 and 30.0 kg/m2 (inclusive), and male subjects were ≥50 kg and female subjects were ≥45 kg;
  3. Meet the diagnostic and Statistical Manual of Mental Disorders (Fifth Edition) (DSM-5) diagnostic criteria for schizophrenia;
  4. The total score of PANSS during screening and baseline was ≤90 points;
  5. Clinical overall impression - severity of disease (CGI-S) score ≤4 points;
  6. Currently not using antipsychotic drugs;
  7. Female subjects of reproductive age, screening and baseline urine pregnancy test results were negative;
  8. Female and male subjects of reproductive age and their spouses agree to use a highly effective contraceptive method during the study medication period and within 3 months after the termination of medication, and no sperm or egg donation is planned;
  9. After fully understanding the purpose, content, process and possible risks of this study, subjects and guardians shall voluntarily participate in this clinical study and sign a written informed consent, and are willing to complete the entire study process according to the requirements of the trial.

Exclusion Criteria:

* Part 1 (SAD) for healthy adults

  1. Other clinically significant diseases;
  2. After C-SSRS assessment, answer "yes" to question 4 or question 5 of the suicidal ideation questionnaire within 1 year, or have a history of suicidal behavior;
  3. allergies to multiple food or drug allergies, or known allergies to test drug ingredients;
  4. Within 2 weeks before the trial (or 5 half-lives of the drug, whichever is longer) or plan to take any medication during the trial, including prescription and over-the-counter drugs, Chinese herbal medicines, but not including vitamins, dietary supplements;
  5. Drug abusers or those who have used soft drugs (e.g., marijuana) within 3 months prior to the trial, or hard drugs (e.g., cocaine, PCP, etc.) within 1 year prior to the trial;
  6. Have a history of alcoholism or consume more than 14 units of alcohol per week in the last 2 weeks (1 unit = 285 mL for beer, 25 mL for spirits, 150 mL for wine);
  7. Smokers who smoked more than 5 cigarettes per day in the 3 months before the test, or could not stop using any tobacco products during the test;
  8. Blood donation or significant blood loss within 3 months before the first dose of the trial drug (≥450mL within 30 days, excluding blood collection at the screening stage), or a blood donation plan during the study period or within 3 months after the last visit;
  9. Those who had undergone surgery within 3 months prior to screening, or planned to undergo surgery during the study period; Or have undergone medical or surgical treatments that permanently alter the absorption, distribution, metabolism, and excretion of oral drugs (such as gastric or intestinal surgery);
  10. Participating in any clinical trial and taking any clinical trial drug within 3 months before the trial;
  11. Difficulty swallowing capsules and other solid preparations;
  12. The female subject is pregnant or breastfeeding, or the serum pregnancy test is positive;
  13. Difficulty in blood collection, unable to tolerate multiple intravenous blood collection and any blood contraindications;
  14. Positive baseline urine drug test, or positive alcohol breath test;
  15. Measured the blood pressure in the recumbent position, and within 3 minutes of changing the position to the upright position compared with the recumbent position, the systolic blood pressure decreased by ≥20mmHg or the diastolic blood pressure decreased by ≥10mmHg;
  16. During screening or baseline, physical examination, vital signs, laboratory examination (blood routine, blood biochemistry, thyroid function, coagulation function, urine routine, serum prolactin, etc.), infectious disease screening, 12-lead electrocardiogram, abdominal B-ultrasound, chest X-ray and other abnormalities, which were judged by the investigator and were clinically significant, should not be included in the trial;
  17. Positive for viral hepatitis (hepatitis B or hepatitis C), AIDS antibody and treponema pallidum antibody during screening;
  18. Any physical or mental illness or condition that, as determined by the study physician, is likely to increase the risk of the trial, interfere with the subject's adherence to the protocol, or interfere with the subject's completion of the trial.
* Part 2 (MAD) for Schizophrenia patients

  1. Meet the DSM-5 diagnostic criteria for other mental disorders, and the researchers judge that it may have an impact on clinical research;
  2. Other diseases or disorders, as determined by the investigator, that are associated with the clinical trial;
  3. After C-SSRS scale assessment, the answer to question 4 or question 5 in the first 6 months of screening was "yes"; Suicide or self-injury within 1 year prior to screening;
  4. According to the judgment of the researchers, the clinical symptoms related to schizophrenia in this episode (such as severe impulsivity, agitation, etc.) may make it difficult for the patients to persist in completing the entire study process, and they are not suitable to participate in this study;
  5. Received electroconvulsive therapy within 3 months before screening;
  6. Use of long-acting antipsychotics within 6 months prior to screening;
  7. A history of epilepsy;
  8. Previous history of malignant syndrome;
  9. The presence of any surgical condition or condition that may significantly affect drug absorption, distribution, metabolism, and excretion, or that may pose a hazard to participants in the trial;
  10. Have a history of severe allergies;
  11. Female subjects were pregnant, puerperal, or lactating at the time of screening or baseline;
  12. Those who have a history of drug abuse within 1 year before screening;
  13. A history of alcohol abuse in the six months prior to screening (i.e. drinking more than 14 standard units per week, 1 standard unit =360 mL beer or 45 mL spirits with 40% alcohol or 150 mL wine), or fail to stop alcohol during the study period;
  14. Smoking more than 5 cigarettes per day (including e-cigarettes) in the 3 months prior to screening, or cannot stop smoking during the study period;
  15. Abnormal physical examination, vital signs, 12-ECG, or lab tests at screening or baseline, which may affect clinical research, as assessed by the study investigator;
  16. Non-negative hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV-Ab), human immunodeficiency virus antibody (HIV-Ab) and syphilis serological test during screening;
  17. Blood donation or blood loss ≥200ml within 1 month before screening;
  18. Participate in any interventional clinical trial within 3 months prior to screening;
  19. Other situations in which the investigator deems it inappropriate to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events(AE) , serious AEs and AE leading to withdrawal from treatment. | SAD: Baseline to Day 6; MAD: Baseline to Day 42
  An AE is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. A serious AE (SAE) is any untoward medical occurrence that at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; or is a congenital anomaly/birth defect.
Changes from baseline in lab tests | SAD: Baseline to Day 6; MAD: Baseline to Day 35
  Laboratory tests include blood routine, urine routine, blood biochemistry, coagulation function and serum prolactin, etc.
Changes from baseline in vital signs | SAD: Baseline to Day 6; MAD: Baseline to Day 35
  Vital signs include blood pressure (BP), pulse rate, respiration and body temperature.
Change from baseline in body weight | SAD: Baseline to Day 6; MAD: Baseline to Day 29
  Body weight was measured in kilograms (Kg).
Change from baseline in Electrocardiogram (ECG) | SAD: Baseline to Day 6; MAD: Baseline to Day 35;
  ECG parameters including heart rate, PR interval, RR interval and QTcF, etc.
Change from Baseline in Columbia - Suicide Severity Rating Scale (C-SSRS) | SAD: Baseline to Day 6; MAD: Baseline to Day 35
  C-SSRS is a scale capturing occurrence, severity, and frequency of suicide-related thoughts and behaviors, and has a binary response (yes/no). Suicidal Ideation: a "yes" answer to any one of 5 suicidal ideation questions: Wish to be Dead, Non-specific Active Suicidal Thoughts, Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act, Active Suicidal Ideation with Some Intent to Act, without Specific Plan, Active Suicidal Ideation with Specific Plan and Intent. Suicidal Behavior: a "yes" answer to any of 5 suicidal behavior questions: Preparatory Acts or Behavior, Aborted Attempt, Interrupted Attempt, Actual Attempt (non-fatal), Completed Suicide.
Change from baseline in Abnormal Involuntary Movement Scale (AIMS) | SAD: Baseline to Day 6; MAD: Baseline to Day 35
  AIMS is a rating scale measuring involuntary movements known as tardive dyskinesia, that sometimes develop as a side effect of long-term treatment with antipsychotic medications. The AIMS score was calculated as the sum of questions 1 through 7 of the AIMS instrument, which includes assessments of involuntary movements in the face, lips, jaw, tongue, upper and lower extremities, and neck/shoulders/hips. Each item is rated on a five-point scale of severity from 0-4 with 0 (none), 1 (minimal), 2 (mild), 3 (moderate), 4 (severe). Total scores range from 0 to 28.
Change from baseline in Barnes Akathisia Rating Scale (BARS) | SAD: Baseline to Day 6; MAD: Baseline to Day 35
  BARS is a rating scale that is administered by physicians to assess the severity of drug-induced akathisia, which is a movement disorder characterized by a feeling of inner restlessness and a compelling need to be in constant motion, as well as by actions such as rocking while standing or sitting, lifting the feet as if marching on the spot, and crossing and uncrossing the legs while sitting. The following subcategories are scored: objective akathisia, subjective awareness of restlessness and subjective distress related to restlessness and are rated on a 4-point scale from 0-3. In addition, the global clinical assessment of akathisia uses a 6-point scale ranging from 0-5. Total score ranges from 0 to 14 with a higher score indicating increased severity.
Change from baseline in Simpson-Angus Scale (SAS) | SAD: Baseline to Day 6; MAD: Baseline to Day 35
  SAS is a 10-item testing instrument used to evaluate drug-related extrapyramidal syndromes. The following items are included in the SAS: gait, arm dropping, shoulder shaking, elbow rigidity, wrist rigidity, leg pendulousness, head dropping, glabella reflex, tremor, and salivation. Total score ranges from 0 to 40 with a higher score indicating increased severity.

SECONDARY OUTCOMES:
Cmax | SAD: up to Day3
  Maximum plasma concentration
Tmax | SAD: up to Day3
  Time to Cmax
AUC0-t | SAD: up to Day3; MAD: up to Day 30
  Area under the plasma concentration-time curve from time 0 to the last of measurable concentration
AUC0-∞ | SAD: up to Day3; MAD: up to Day 30
  Area under the plasma concentration-time curve from 0 to infinity
λz | SAD: up to Day3
  terminal rate constant
t½ | SAD: up to Day3; MAD: up to Day 30
  elimination half-life
CL/F | SAD: up to Day3
  apparent plasma clearance
Vd/F | SAD: up to Day3
  apparent volume of distribution
MRT | SAD: up to Day3
  mean residence time
Css, max | MAD: up to Day 30
  Maximum concentration at steady state
Css, min | MAD: up to Day 30
  Minimum concentration at steady state
Css, av | MAD: up to Day 30
  Average concentration at steady state
Tss, max | MAD: up to Day 30
  Time of the maximum concentration at steady state
AUCss | MAD: up to Day 30
  Area under the concentration-time curve at steady state
Change from Baseline in Positive and Negative Syndrome Scale (PANSS) | MAD: Baseline to Day 35
  PANSS is a 30-item rating scale specifically developed to asses both the positive and negative symptom syndromes of patients with schizophrenia. PANSS is comprised of 30 items and 3 subscales (Positive, Negative, General Psychopathology). An anchored Likert scale from 1 - 7, where values of 2 and above indicate the presence of progressively more severe symptoms, is used to score each item. Individual items are then summed to determine scores for the 3 subscales, as well as a total score. PANSS Positive subscale score range: 7-49. PANSS Negative subscale score range: 7-49. PANSS General Psychopathology subscale score range: 16-112. PANSS total score range: 30-210. Higher PANSS total score means more severe outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojiao Li, Dr., Principal Investigator — The First Hospital of Jilin University
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China